CLINICAL TRIAL: NCT06743789
Title: Dose De-escalation Randomized Phase I/II Trial in Arrhythmia Radioablation for Ventricular Tachycardia: Single Fraction vs Three Fractions
Brief Title: Trial in Arrhythmia Radioablation for Ventricular Tachycardia: Single Fraction vs Three Fractions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-09026474
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: If participants are randomized to either Arm 1 or Arm 2, participants will be in one of the three groups. Each group will enroll 3 participants, based on a criteria of consecutive enrollment over time. After 6 weeks from the last treated participant in Group 1, there will be a review of safety and efficacy of the study intervention in the treated participants before enrolling participants in the next group. This review will continue until the 3rd participant in Group 3 is enrolled and treated. Subsequently the protocol will then move into the follow up phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- 20 Gy Radiation Dose (Arm 1 Group 1) (Experimental): Arm 1:
  Group 1 (3 participants) - will receive a dose of 20 Gy ("Gray", a measurement of radiation) in a single study intervention (one study intervention day)
  Interventions: Radiation: Radiation Therapy
- 15 Gy Radiation Dose (Arm 1 Group 2) (Experimental): Arm 1:
  Group 2 (3 participants) - will receive a dose of 15 Gy in a single study intervention (one study intervention day)
  Interventions: Radiation: Radiation Therapy
- 10 Gy Radiation Dose (Arm 1 Group 3) (Experimental): Arm 1:
  Group 3 (3 participants) - will receive a dose of 10 Gy in a single study intervention (one study intervention day)
  Interventions: Radiation: Radiation Therapy
- 12 Gy Radiation Dose for 3 fractions (Arm 2 Group 1) (Experimental): Arm 2:
  Group 1 (3 participants) - will receive a dose of 12 Gy ("Gray", a measurement of radiation) given over 3 days (Days 1, 2 and 3). (Total radiation dose = 36Gy)
  Interventions: Radiation: Radiation Therapy
- 10 Gy Radiation Dose for 3 fractions (Arm 2 Group 2) (Experimental): Arm 2:
  Group 2 (3 participants) - will receive a dose of 10 Gy ("Gray", a measurement of radiation) given over 3 days (Days 1, 2 and 3). (Total radiation dose = 30Gy)
  Interventions: Radiation: Radiation Therapy
- 8Gy Radiation Dose for 3 fractions (Arm 2 Group 3) (Experimental): Arm 2:
  Group 3 (3 participants) - will receive a dose of 8 Gy ("Gray", a measurement of radiation) given over 3 days (Days 1, 2 and 3). (Total radiation dose = 24Gy)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Group 1 (3 participants) - will receive a dose of 20 Gy ("Gray", a measurement of radiation) in a single study intervention (one study intervention day)
  Other Names: Cardio Ablation
  Arms: 20 Gy Radiation Dose (Arm 1 Group 1)
Radiation: Radiation Therapy — Group 2 (3 participants) - will receive a dose of 15 Gy in a single study intervention (one study intervention day)
  Other Names: Cardio Ablation
  Arms: 15 Gy Radiation Dose (Arm 1 Group 2)
Radiation: Radiation Therapy — Group 3 (3 participants) - will receive a dose of 10 Gy in a single study intervention (one study intervention day)
  Other Names: Cardio Ablation
  Arms: 10 Gy Radiation Dose (Arm 1 Group 3)
Radiation: Radiation Therapy — Group 1 (3 participants) - will receive a dose of 12 Gy given over 3 days (Days 1, 2 and 3). (Total radiation dose = 36Gy)
  Other Names: Cardio Ablation
  Arms: 12 Gy Radiation Dose for 3 fractions (Arm 2 Group 1)
Radiation: Radiation Therapy — Group 2 (3 participants) - will receive a dose of 10 Gy given over 3 days (Days 1, 2 and 3). (Total radiation dose = 30Gy)
  Other Names: Cardio Ablation
  Arms: 10 Gy Radiation Dose for 3 fractions (Arm 2 Group 2)
Radiation: Radiation Therapy — Group 3 (3 participants) - will receive a dose of 8 Gy given over 3 days (Days 1, 2 and 3). (Total radiation dose = 24Gy)
  Other Names: Cardio Ablation
  Arms: 8Gy Radiation Dose for 3 fractions (Arm 2 Group 3)

SUMMARY:
This is a research study that aims to understand if giving a lower dose of treatment all at once is as effective and safe as dividing it into three smaller doses for patients with a heart condition called refractory ventricular tachycardia (VT). These patients have not exhibited positive responses to conventional medications or procedures. This study aims to explore whether an alternative approach could yield more beneficial outcomes.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) is a life-threatening heart rhythm disorder that arises from areas of diseased tissue in the heart. Treatment of VT can involve anti-arrhythmic drugs and catheter-based ablations. Unfortunately, despite multiple antiarrhythmic drugs, as well as the catheter-based ablation procedures, VT continues to persist in your case. At this point in time, The investigators believe that stereotactic body radiotherapy (SBRT) remains the only possible option to potentially treat VT. The investigators hypothesize that by administering SBRT at different dose levels and fractionation may achieve a better therapeutic ratio, defined as comparable efficacy with less risk of toxicity due to lower dose exposure to the normal tissue, including the heart vasculature, in patients when compared to VT patients who receive a dose of 25Gy in a single fraction which is the current treatment option.

This is a randomized dose de-escalation trial where the patients will be randomized in in one of the two experimental arms, receiving 1 single fraction OR 3 daily consecutive fractions of RT, and will be treated into a prespecified dose level group, based on the study development. The study includes three de-escalated consecutive dose level groups for each of two randomized treatment arms and there will be 3 patients per group and each group will receive a particular radiation treatment either as single treatments or three treatments.

The purpose of this treatment is to safely reduce episodes of VT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Structural heart disease:

  1. Ischemic cardiomyopathy
  2. Non-ischemic cardiomyopathy
  3. Hypertrophic cardiomyopathy
* Refractory VT severity:

  1. VT leading to ICD shock with minimum 3 episodes in any 3-month period without reversible cause;
  2. Failed or intolerant to antiarrhythmic drug therapy (either amiodarone or ≥ 2 AADs) AND failed ablation (CA)
  3. OR ablation (CA) contraindicated
* Ability to understand study protocol and to write informed consent
* Willing to comply with specified pre-, post- and follow-up testing, evaluations and requirements
* Expected to remain available for at least 36 months after enrollment

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Prior chest radiation therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by number of subjects with a reduction ≥ 60% (tracked by ICD recordings) ventricular tachycardia (VT) episodes | 6 months before treatment
Efficacy as measured by number of subjects with a reduction ≥ 60% (tracked by ICD recordings) ventricular tachycardia (VT) episodes | 6 weeks post treatment
Number of treatment-related serious adverse events (SAEs) | 6 weeks post treatment
  Safety: SAEs rate ≤ 30% defined using Common Terminology Criteria for Adverse Events (CTCAE) criteria (version 5.0) that could be treatment-related (possibly, probably, or definitely related to treatment) at 6 weeks after treatment is considered clinically acceptable.
  The SAEs are defined as any grade 3 toxicity requiring hospitalization or any grade 4 to 5 toxicity.

SECONDARY OUTCOMES:
Number of ventricular tachycardia (VT) episodes | 3 months post
Number of ventricular tachycardia (VT) episodes | 6 months post
Number of ventricular tachycardia (VT) episodes | 12 months
Number of subacute treatment side-effects | 3 months post
  Subacute treatment side effects, defined as any grade according to CTCAE criteria (version 5.0)
Number of subacute treatment side-effects | 6 months post
  Subacute treatment side effects, defined as any grade according to CTCAE criteria (version 5.0)
Number of late Adverse events | 1 year post
  Long term treatment side effects, defined as any grade according to CTCAE criteria (version 5.0)
Number of late Adverse events | 2 year post
  Long term treatment side effects, defined as any grade according to CTCAE criteria (version 5.0)
Overall survival | 1 year post
  Overall survival, defined as time calculated from treatment to death for any cause;
Overall survival | 2 year post
  Overall survival, defined as time calculated from treatment to death for any cause;
Recurrence free survival | 3 months post
  Recurrence free survival, defined as "time to VT storm" with VT storm defined as ≥ 3 VT/VF episodes leading to ICD therapy within 24 hours
Recurrence free survival | 6 months post
  Recurrence free survival, defined as "time to VT storm" with VT storm defined as ≥ 3 VT/VF episodes leading to ICD therapy within 24 hours
Recurrence free survival | 12 months post
  Recurrence free survival, defined as "time to VT storm" with VT storm defined as ≥ 3 VT/VF episodes leading to ICD therapy within 24 hours
Recurrence free survival | 24 months post
  Recurrence free survival, defined as "time to VT storm" with VT storm defined as ≥ 3 VT/VF episodes leading to ICD therapy within 24 hours
Number of incidents of implantable cardiac device (ICD) shock | 3 months before treatment
Number of incidents of implantable cardiac device (ICD) shock | 3 months post treatment
Number of Anti-Arrhythmic Drugs (AADs) administration | 3 months before treatment
  Any reduction in Anti-Arrhythmic Drugs (AADs) administration
Number of Anti-Arrhythmic Drugs (AADs) administration | 3 months post treatment
  Any reduction in Anti-Arrhythmic Drugs (AADs) administration

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No